CLINICAL TRIAL: NCT00667511
Title: Comparison of Nocturnal Hemodialysis (NHD) and Short Daily Hemodialysis (DHD) With the NxStage® System One™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NxStage Medical (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP0010
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Kidney Failure, Chronic; End-Stage Renal Disease
Keywords: ESRD; End Stage Renal Disease; Daily Hemodialysis; Nocturnal Hemodialysis; Hemodialysis; Kidney Failure; Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home Short Daily Hemodialysis (Active Comparator): Intervention: Patients perform short daily hemodialysis (2 to 4 hour treatments) in the home setting using the NxStage System One.
  Interventions: Device: NxStage System One
- Home Nocturnal Hemodialysis (Experimental): Intervention: Patients perform nocturnal hemodialysis (6 to 10 hour treatments) in the home setting using the NxStage System One.
  Interventions: Device: NxStage System One

INTERVENTIONS:
Device: NxStage System One — Comparison of Nocturnal (NHD) and Short Daily Hemodialysis (DHD) with the NxStage System One

SUMMARY:
The purpose of this study is to determine whether or not nocturnal hemodialysis is equivalent to short daily hemodialysis on a per treatment basis, using the NxStage System One in the home setting.

DETAILED DESCRIPTION:
End Stage Renal Disease (ESRD) continues to be a devastating clinical condition. The number of patients in 2004 affected by ESRD in the United States rose to 472,000. More than 104,000 new patients began therapy for ESRD in 2004 (1.5% greater than in 2003), while the prevalent dialysis population reached nearly 336,000 (3.4% higher). Total Medicare costs for ESRD in 2004 rose to $20.1 billion while non-Medicare costs rose to $12.4 Billion(1).

Treatment options for ESRD patients are currently limited to either transplantation or dialysis. As daily hemodialysis (DHD) continues to gain widespread acceptance in the dialysis community, there is also renewed interest in nocturnal hemodialysis (NHD) therapy.

NHD has the potential to provide certain advantages over both DHD and conventional thrice-weekly in-center HD. NHD typically consists of 6 - 10 hour treatments while the patient sleeps, providing more gentle fluid removal, more time for equilibration, improved hemodynamic stability and superior clearance of larger solutes(2).

The proposed study plans to explore whether or not NHD is equivalent to DHD on a per treatment basis, using the NxStage System One in the home setting.

1. United States Renal Data System 2006 Annual Data Report: Atlas of End-Stage Renal Disease in the United States, NIH, NIDDK, Bethesda, MD, 2006
2. Lacson E, Diaz-Buxo J: Daily and Nocturnal Hemodialysis: How do they stack up? American Journal Kidney Disease, Vol 38(2) Aug 2001: 225-239.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a stable prescription in the short daily home environment using the NxStage System One prior to enrollment.

Exclusion Criteria:

* Patients are not eligible if:

  * they are currently enrolled in another drug or device study which could impact the successful completion of this study
  * they are currently on NHD, or less than 3 months since discontinuing NHD
  * if they were previously enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kravitz, Study Director — NxStage Medical
Locations (9):
- United States (9):
  - Satellite Healthcare/Wellbound, San Jose, California
  - Circle Medical Management, Chicago, Illinois
  - Indiana University Dialysis Center, Indianapolis, Indiana
  - Kansas Nephrology Research Institute, LLC, Wichita, Kansas
  - Barnes Jewish Dialysis Center, St Louis, Missouri
  - Dialysis Center of Lincoln, Lincoln, Nebraska
  - Rubin Dialysis, Saratoga Springs, New York
  - DaVita Grapevine at Home, Grapevine, Texas
  - DaVita Bluemound Home Dialysis, Wauwatosa, Wisconsin

REFERENCES:
- [Derived] Liu F, Abra G, Gupta N, Schiller B, Rivara MB. How I Treat Nocturnal Home Hemodialysis-An Underprescribed but Essential Home Dialysis Modality in the United States. Clin J Am Soc Nephrol. 2025 Oct 10. doi: 10.2215/CJN.0000000927. Online ahead of print. No abstract available. PMID 41071621

RESULTS

PARTICIPANT FLOW:
Groups:
- Home Short Daily Hemodialysis Then Home Nocturnal Hemodialysis: Intervention 1: Patients performed short daily hemodialysis (DHD) (2 to 4 hour treatments) in the home setting using the NxStage System One for an 8 week period.
  Intervention 2: Patients completing Intervention 1 and successfully completing a 4 week training/transition period proceeded to perform nocturnal hemodialysis (NHD) (6 to 10 hour treatments) in the home setting using the NxStage System One for an 8 week period.
  In this prospective, two treatment, cross-over study, 58 End Stage Renal Disease patients >18 years of age who were currently stable on home DHD were enrolled. Enrolled patients performed Intervention 1 as the first phase of the cross-over study. Fifty-one patients completed Intervention 1 and seven patients dropped out. Forty-three patients completed the training/transition period and performed Intervention 2 as the second phase of the cross-over study. Thirty-nine patients completed Intervention 2 and four patients dropped out.
Period: Intervention 1: Home DHD
Arm/Group | Home Short Daily Hemodialysis Then Home Nocturnal Hemodialysis
Started | 58
Completed | 51
Not Completed | 7
Period: Training/Transition Period
Arm/Group | Home Short Daily Hemodialysis Then Home Nocturnal Hemodialysis
Started | 51
Completed | 43
Not Completed | 8
Period: Intervention 2: Home NHD
Arm/Group | Home Short Daily Hemodialysis Then Home Nocturnal Hemodialysis
Started | 43
Completed | 39
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: 58 patients were enrolled in the cross-over study. Patients were required to complete the home short daily hemodialysis phase before transitioning to the home nocturnal hemodialysis phase.
Groups:
- Home Short Daily Hemodialysis Then Home Nocturnal Hemodialysis: Intervention 1: Patients performed short daily hemodialysis (DHD) (2 to 4 hour treatments) in the home setting using the NxStage System One for an 8 week period.
  Intervention 2: Patients completing Intervention 1 and successfully completing a 4 week training/transition period proceeded to perform nocturnal hemodialysis (NHD) (6 to 10 hour treatments) in the home setting using the NxStage System One for an 8 week period.
Arm/Group | Home Short Daily Hemodialysis Then Home Nocturnal Hemodialysis
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy: Compare the Ability to Deliver the Clinically Prescribed Amount of Therapy in the Nocturnal Hemodialysis and Short Daily Hemodialysis Phases.
Description: The primary efficacy endpoint for the study was the ability to deliver the clinically prescribed amount of therapy, defined by attainment of a delivered volume that was at least 90% of the prescribed volume (10% difference in success rate is the upper boundary of the 95% confidence interval).
Time Frame: Study Week 20
Population: Includes all electronically captured treatments.
Measure: Number (95% Confidence Interval); unit: percentage of successful treatments
Units Other Than Participants: Treatments
Groups:
- Home Short Daily Hemodialysis: Intervention 1: Patients perform short daily hemodialysis (2 to 4 hour treatments) in the home setting using the NxStage System One.
- Home Nocturnal Hemodialysis: Intervention 2: Patients perform nocturnal hemodialysis (6 to 10 hour treatments) in the home setting using the NxStage System One.
Arm/Group | Home Short Daily Hemodialysis | Home Nocturnal Hemodialysis
Number analyzed (Participants) | 58 | 43
Number analyzed (Treatments) | 1866 | 1431
percentage of successful treatments | 90.9 [89.2 to 92.6] | 91.7 [89.9 to 93.5]

2. Primary Outcome: Primary Safety: Compare the Composite Intradialytic and Interdialytic Adverse Event Profile in the Nocturnal Hemodialysis and Short Daily Hemodialysis Phases.
Description: The primary safety endpoint for the study was the composite intradialytic and interdialytic adverse event (AE) profile.
Time Frame: Study Week 20
Population: Includes all patient reported treatments.
Measure: Number; unit: events per 100 treatments
Units Other Than Participants: Treatments
Arm/Group | Home Short Daily Hemodialysis | Home Nocturnal Hemodialysis
Number analyzed (Participants) | 58 | 43
Number analyzed (Treatments) | 2373 | 1792
events per 100 treatments | 8.3 | 6.9

ADVERSE EVENTS:
Time Frame: Adverse events were reported during the 20 week period of study participation.
Groups:
- Nocturnal Home Hemodialysis: Intervention 2: Patients perform nocturnal hemodialysis (6 to 10 hour treatments) in the home setting using the NxStage System One.
Arm/Group | Home Short Daily Hemodialysis | Nocturnal Home Hemodialysis
Serious Adverse Events (participants affected / at risk) | 13/58 | 5/43
Other Adverse Events (participants affected / at risk) | 40/58 | 30/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home Short Daily Hemodialysis (N=58) | Nocturnal Home Hemodialysis (N=43)
Angina/Chest Pain (Cardiac disorders) | 2 (2) | 0 (0)
Musculoskeletal Injuries (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) — Non-dialysis related joint sprains, tears, and fractures
Hypertension (Renal and urinary disorders) | 1 (1) | 0 (0)
Vascular Access Issues (Vascular disorders) | 4 (6) | 1 (2)
Infection (General disorders) | 2 (2) | 2 (2)
Abdominal Pain (General disorders) | 1 (2) | 0 (0)
Cerebrovascular Accident (Vascular disorders) | 1 (1) | 0 (0)
Eye surgery (Surgical and medical procedures) | 0 (0) | 1 (1) — non-dialysis related
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home Short Daily Hemodialysis (N=58) | Nocturnal Home Hemodialysis (N=43)
Cold/Flu-like Symptoms (General disorders) | 12 (17) | 6 (8)
Other (General disorders) | 9 (26) | 4 (20) — other singular non-dialysis-related events
Clotted Dialysis Blood Lines (General disorders) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 5 (8)
Vascular Access Problems (Vascular disorders) | 12 (20) | 8 (16) — i.e. poor access flow, painful access, bleeding
Hypotension/Hypovolemia/Cramping (Renal and urinary disorders) | 22 (71) | 13 (26)
Dialysis-related blood loss (Renal and urinary disorders) | 5 (6) | 3 (5)
Fatigue (General disorders) | 3 (4) | 4 (5)
General Bodily Pain (General disorders) | 2 (4) | 3 (4) — i.e. shoulder pain, back pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days